CLINICAL TRIAL: NCT04394910
Title: Impact of Antioxidant Juice Intake on Brain Injury and Placental Pathology in Infants With Intrauterine Growth Restriction (IUGR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of California, Los Angeles (Other); POM Wonderful LLC (Industry)
Responsible Party: Principal Investigator, Terrie Inder, Chair, Department of Pediatric Newborn Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014P000870
Record Dates: First submitted 2020-05-11; First posted 2020-05-20 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pomegranate Juice (Experimental): Dietary supplementation with 8 oz. commercially-available pomegranate juice consumed daily.
  Interventions: Dietary Supplement: Pomegranate Juice
- Placebo Juice (Placebo Comparator): Dietary supplementation with 8 oz. placebo juice (identical to pomegranate juice but lacking polyphenols) consumed daily.
  Interventions: Dietary Supplement: Placebo Juice

INTERVENTIONS:
Dietary Supplement: Pomegranate Juice
  Arms: Pomegranate Juice
Dietary Supplement: Placebo Juice
  Arms: Placebo Juice

SUMMARY:
Infants diagnosed with intrauterine growth restriction are at increased risk for brain injury in the neonatal period, and eventually increased risk for adverse long-term neurodevelopmental outcomes. This kind of growth restriction is often caused by long-term placental insufficiency leading to chronic lack of oxygen in the brain during development. Pomegranate juice is one of the highest polyphenol-containing dietary supplements commercially available. Previous studies have shown that pomegranate-derived polyphenols are potent neuroprotective antioxidants with no proven side effects. The investigators hypothesize that maternal dietary supplementation with pomegranate juice during the last trimester of pregnancy will reduce the effects of exogenous stimuli contributing to placental insufficiency, and will enhance brain growth and development in the IUGR population.

DETAILED DESCRIPTION:
The current study seeks to investigate the impact of maternal dietary supplementation with pomegranate juice on placental morphology and on subsequent newborn brain development and function. A total of 99 consenting women carrying fetuses with a diagnosis of intrauterine growth restriction (IUGR) in the third trimester were randomized to one of two arms.

Treatment Group: Expecting mothers in this group will be randomized to consume 8oz of pomegranate juice daily. Participants will keep a daily diary documenting compliance with the regimen. Participants will continue daily intake until delivery.

Placebo group: Expecting mothers will be randomized to consume an 8oz of pomegranate free juice placebo that matches taste, calories, and appearance to regular pomegranate juice but lacks polyphenols. Participants will keep a diary of daily intake to help ensure compliance similar to the treatment group. Participants will continue to placebo until delivery.

Both groups: Maternal blood and urine samples will be collected prior to starting the juice regimen in order to establish baseline metabolite status. For the first 84 mothers enrolled, a fetal MRI was scheduled prior to beginning the juice regimen. Phase I participants will undergo two fetal echocardiograms: one before starting the juice regimen, and a second two weeks into the juice regimen to establish the safety of high polyphenol intake on fetal heart development. All women will be contacted on a weekly basis to assess compliance. At the time of delivery, maternal blood and urine, and cord blood will be collected and sent for analysis to test for the presence of dimethylellagic acid glucuronide (DMEAG) and urolithin A glucuronide (UAG), polyphenic components of pomegranate juice. Placental material will be sent for formal pathological exam.

If clinically stable, MRI will be undertaken without sedation at term equivalent (38-41 weeks CGA). Infants will undergo testing of cognitive, gross and fine motor, and speech skills at around 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

- Expecting mother with a fetal diagnosis of less than 5th percentile on the Doubilet fetal growth curve

Exclusion Criteria:

* Multiple congenital abnormalities
* Known fetal chromosomal disorder
* Maternal illicit drug or alcohol intake

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2016-01-16 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-26 (Actual)

PRIMARY OUTCOMES:
Infant brain injury assessed on term-equivalent brain magnetic resonance image (MRI) using the Kidokoro injury scoring system. | One time occurrence at birth or term-equivalent age if infant is born preterm.
  The Kidokoro scale is a comprehensive, objective scoring system for classifying the nature and extent of neonatal brain injury on MRI (Kidokoro et al. American Journal of Neuroradiology. 2013; 34(11):2208-14).
Total and regional infant brain volumes assessed on term equivalent brain MRI using MANTiS. | One time occurrence at birth or term-equivalent age if infant is born preterm.
  MANTiS (Morphologically Adaptive Neonatal Tissue Segmentation) describes neonate-specific brain tissue segmentation into 8 categories using Statistical Parametric Mapping (SPM) software (Beare et al. Frontiers in Neuroinformatics. 2016;10:12).
Diffusion tensor imaging measures of fractional anisotropy (FA), and mean (MD), radial (RD), and axial (AD) diffusivity from infant term equivalent brain MRI. | One time occurrence at birth or term-equivalent age if infant is born preterm.
  FA, MD, RD, and AD will be measured from a diffusion-weighted sequence on brain MRI.

SECONDARY OUTCOMES:
Cognitive, motor, and language neurodevelopment scores on the Bayley III exam. | The Bayley III exam will be administered at a one-time visit scheduled between 18-36 months.
  The Bayley Scores of Infant and Toddler Development (Edition III) is a comprehensive examination tool used to assess neurodevelopment in infants and toddlers up to 42 months.
Maternal compliance with juice regimen. | Comparison of one pre-juice regimen UA and DMEAG concentration measurement (ng/mL) to one post-juice regimen blood and urine concentration measurement (ng/mL) collected at the time of delivery.
  Maternal compliance with the assigned juice regimen is assessed by participant logbook record and assessment of change in polyphenols (urolithin A and dimethylellagic glucuronide concentration, ng/mL) in maternal urine and blood at enrollment and in maternal urine, blood and cord blood at the time of delivery.

OTHER OUTCOMES:
Placental weight. | The placenta will be weighed as part of routine pathology exam within 1-3 days of delivery.
  Weight of the placenta measured in grams.
Incidence of pre-eclampsia. | The electronic medical record will be reviewed within 1 week of delivery.
  Incidence of pre-eclampsia requiring medication as documented in the medical record.
Gestational age at delivery. | The electronic medical record will be reviewed within 1 week of delivery.
  Gestational age at delivery based on ultrasound dating acquired at less than 12 weeks' gestation as documented in the medical record.
Incidence of resuscitation at delivery. | The electronic medical record will be reviewed within 1 week of delivery.
  Incidence of infant resuscitation at delivery measured by APGAR scores assigned at birth and documented in the medical record.
Cord gas characteristics. | The electronic medical record will be reviewed within 1 week of delivery.
  Umbilical artery cord gas pH and base deficit as documented in the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Terrie E Inder, MD, MBChB, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) cannot be shared publicly because the investigators had not previously sought Institutional Review Board (IRB) approval for public sharing of participant data as part of the informed consent process. However, the investigators will gladly share with any investigator the de-identified minimal raw data set needed to replicate the study upon request.

REFERENCES:
- [Derived] Ross MM, Cherkerzian S, Mikulis ND, Turner D, Robinson J, Inder TE, Matthews LG. A randomized controlled trial investigating the impact of maternal dietary supplementation with pomegranate juice on brain injury in infants with IUGR. Sci Rep. 2021 Feb 11;11(1):3569. doi: 10.1038/s41598-021-82144-0. PMID 33574371